CLINICAL TRIAL: NCT06119464
Title: Re-Purposing the Ordering of 'Routine' Laboratory Tests in Hospitalized Medical Patients (RePORT Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other); University of British Columbia (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Anshula Ambasta, Clinical Assistant Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: REB17-1215
Record Dates: First submitted 2023-10-26; First posted 2023-11-07 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Utilization, Health Care
Keywords: Overutilization of lab test; Multimodal intervention; Lab test overuse; Laboratory; Hospital
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial, randomizing the sequence of entry into intervention at a cluster level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unexposed to intervention (control period) (No Intervention): This is the time period of the study where hospital clusters are not receiving the intervention
- Exposed to intervention (intervention period) (Experimental): This is the time period of the study where hospital clusters are receiving the multimodal intervention.
  Interventions: Other: Multimodal Intervention: Education; Other: Multimodal Intervention: Audit and Feedback; Other: Multimodal Intervention: Patient Engagement; Other: Multimodal Intervention: System Changes

INTERVENTIONS:
Other: Multimodal Intervention: Education — The multimodal intervention bundle consists of education, audit and feedback, patient engagement, and system changes.
  Arms: Exposed to intervention (intervention period)
Other: Multimodal Intervention: Audit and Feedback — The multimodal intervention bundle consists of education, audit and feedback, patient engagement, and system changes.
  Arms: Exposed to intervention (intervention period)
Other: Multimodal Intervention: Patient Engagement — The multimodal intervention bundle consists of education, audit and feedback, patient engagement, and system changes.
  Arms: Exposed to intervention (intervention period)
Other: Multimodal Intervention: System Changes — The multimodal intervention bundle consists of education, audit and feedback, patient engagement, and system changes.
  Arms: Exposed to intervention (intervention period)

SUMMARY:
Laboratory test overuse occurs when tests are ordered repetitively, without due consideration of impact on clinical status. Repetitive inpatient lab testing often provides limited value for patient outcomes while increasing healthcare costs, patient discomfort, and unnecessary transfusions and prolonging hospitalizations. The research study aims to reduce laboratory test overuse in hospitals through implementation of a comprehensive, multi-disciplinary, and multi-faceted intervention bundle that includes audit and feedback reports, clinician education, clinical decision support tool, and patient infographics across 14 hospitals in Alberta.

DETAILED DESCRIPTION:
Background: Laboratory and Pathology testing contributes to rising health care expenditure. A relatively large percentage (up to 42%) of laboratory testing can be considered wasteful. Redundant testing alone has been estimated to waste up to 5 billion dollars annually in the United States of America. Laboratory over-utilization leads to false positives that promotes further inappropriate testing and procedures, interruption of normal sleep pattern of inpatients, as well as iatrogenic anemia and pain. A Canadian study showed significant hemoglobin reductions as a result of phlebotomy. Studies support the safe reduction of repetitive laboratory testing without negative effects on adverse events, readmission rates, critical care utilization, or mortality.

The aim of this research study is the following:

1. To implement a multimodal intervention bundle containing healthcare provider and patient engagement tools for hospitalized medical inpatients in 14 hospitals across the province of Alberta in Canada using a cluster randomized stepped-wedge design
2. To evaluate the impact of the intervention bundle on laboratory test utilization of six target laboratory tests (complete blood count, electrolytes, creatinine, urea, partial thromboplastin time, and international normalized ratio), costs, and patient safety outcomes.

This intervention bundle will be implemented across all the adult hospital sites in Alberta starting January 2023 and evaluated until October 2024.

ELIGIBILITY:
Inclusion Criteria:

* all participants (patients and healthcare providers) within enrolled adult hospitals in Alberta of medical and hospitalist units during study period

Exclusion Criteria:

* outside of the above-mentioned province
* hospitals not enrolled
* non-medical units (eg. ICU, surgical, pediatric, obstetrical units)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251817 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of routine laboratory tests ordered per patient-day in the intervention versus control periods | 1 year 9 months
  Number of the six target laboratory tests (complete blood count, electrolytes, creatinine, urea, international normalized ratio and partial thromboplastin time) ordered per patient-day

SECONDARY OUTCOMES:
Costs associated with routine and all common laboratory test ordered | 1 year 9 months
  Costs of test and associated costs with and without intervention
Proportion of hospital patient lab-free days | 1 year 9 months
  Number of hospital patient-days not associated with laboratory blood draws
Proportion of critically abnormal test results | 1 year 9 months
  As defined by lab standards, we will track the proportion of critically abnormal test results
Length of stay | 1 year 9 months
  Patient length of stay on the unit
Transfer to Intensive Care Unit | 1 year 9 months
  Transfer rate to Intensive Care Unit
In-patient and 30-day patient mortality over study period | 30 days post discharge
  Mortality rate in hospital and at 30-days post discharge
30-day post discharge readmission rate | 30 days post discharge
  Hospital re-admission within 30 days post discharge
Number of all common laboratory tests | 1 year 9 months
  Number of all common laboratory tests (tests that contribute to >80% of hospital laboratory test utilization during study period) per patient-day.

CONTACTS AND LOCATIONS:
Overall Officials: Anshula Ambasta, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Study data and results will be available for sharing with other researchers who follow the ethical and institutional protocols required by hospitals and health systems involved to obtain the same data